CLINICAL TRIAL: NCT06958367
Title: Effect of Dexmedetomidine on Acute Kidney Injury After Ascending Aortic Surgeries: Placebo-controlled, Randomised Controlled Trial
Brief Title: Effect of Dexmedetomidine on Acute Kidney Injury After Ascending Aortic Surgeries
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU MD43/2025
Record Dates: First submitted 2025-04-06; First posted 2025-05-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Aki After Ascending Aortic Surgeries
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active arm (Active Comparator): Group (A): will receive Dexmedetomidine which will be mixed with 0.9% saline to achieve a concentration of 4ug/ml which will be continuously infused at a rate of 0.4 ug/kg/hr for 24 hours starting immediately after anesthetic induction
  Interventions: Drug: Dexmedetomidine
- control arm (Placebo Comparator): Group (B): the control group will receive an infusion of an equivalent volume of a 0.9% saline for the same duration
  Interventions: Drug: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Dexmedetomidine — the effect of dexmedetomidine administration on AKI after ascending aortic surgeries requiring CPB in a placebo-controlled randomised controlled trial.
  Arms: active arm
Drug: Normal Saline (Placebo) — Group (B): the control group will receive an infusion of an equivalent volume of a 0.9% saline for the same duration
  Arms: control arm

SUMMARY:
Acute kidney injury (AKI) is a frequent and serious complication after ascending aortic surgeries requiring cardiopulmonary bypass (CPB). Dexmedetomidine, a selective α-2 adrenoreceptor agonist, may reduce AKI because of its sympatholytic and anti-inflammatory effects against ischaemia reperfusion injury. We investigate the effect of dexmedetomidine administration on AKI after ascending aortic surgeries requiring CPB in a placebo-controlled randomised controlled trial.

DETAILED DESCRIPTION:
The aim of the study is the effect of dexmedetomidine administration on AKI after ascending aortic surgeries requiring CPB in a placebo-controlled randomised controlled trial.

Type of Study: A prospective, randomized, comparative, single-center, double-blinded, interventional clinical trial study.

Study Setting: Cardiac Intensive care, Cardiac Surgical Academy Faculty of Medicine - Ain Shams University, Cairo, Egypt.

Study Period: 1 year after approval of the ethical committee of the faculty of medicine, Ain Shams University.

Study Population: 78 patients will be endorsed as follows:

1. Group (A): will receive Dexmedetomidine which will be mixed with 0.9% saline to achieve a concentration of 4ug/ml which will be continuously infused at a rate of 0.4 ug/kg/hr for 24 hours starting immediately after anesthetic induction
2. Group (B): the control group will receive an infusion of an equivalent volume of a 0.9% saline for the same duration

Inclusion Criteria:

* Age: 20-70 yrs
* Scheduled for aortic surgery under CPB

Exclusion Criteria:

* Patient refusal to participate
* Congestive heart failure with a left ventricular ejection fraction <45%
* Uncontrolled arrhythmia combined with unstable hemodynamics
* Acute coronary syndrome.
* Preoperative elevated kidney function (serum urea and serum creatinine).
* Use of ventricular assist devices. Sampling Method: Simple random sampling Sample Size: Sample size was calculated using G*Power software version 3.1.9.2 program, setting the type-1 error (α) at 0.05 and the power (1-β) at 0.9. Result from previous study showed that the incidence of AKI was 13% among cases in dexmedetomidine group, compared to 54% among control group as reported by . Calculation according to these values produced a sample size of 38 cases per group (78 total) with an estimated drop-out rate of 20%.

Ethical Considerations: The procedure will be done under the supervision of the main supervisor. The study will be performed after approval from the Research Ethical Committee (REC), Faculty of Medicine, Ain Shams University. Informed and written consent will be obtained from all participants before starting the study. The study protocol will be explained to the participants before taking their consent to participate in the study.

Study Tools:

All the used interventional medications are approved by the Food and Drug Administration (FDA) and the Pharmacy and Therapeutics Committee (PTC) of Ain Shams University Hospitals.

Dexmedetomidine Hydrochloride: PrecedexR 200 µg/2ml vial , Pfizer, Egypt.

Study Procedures and Intervention:

Consented and enrolled 78 patients will be randomly assigned to one of the following 2 groups:

1. Group (A): will receive Dexmedetomidine which will be mixed with 0.9% saline to achieve a concentration of 4ug/ml which will be continuously infused at a rate of 0.4 ug/kg/hr for 24 hours starting immediately after anesthetic inducion
2. Group (B): the control group will receive an infusion of an equivalent volume of a 0.9% saline for the same duration

A.Preoperative settings:

All patients will be fasting for 8 hours. All patients will have their medical and anesthetic history taken with a full physical examination. Revision of radiological images (ECHO, Carotid Duplex, LL Arterial duplex and Coronary angiography) and routine investigations including CBC, coagulation profile, electrolytes, kidney, and liver profiles will be done.

B.Intraoperative settings:

All subjects will receive institutionally standardised anaesthetic care and CPB management according to our institutional protocol.

Standard monitoring with electrocardiogram (ECG) for heart rate (beats/min), pulse oximetry for (SpO2 as a percentage),trans-oesophageal echocardiography, and invasive monitoring, including radial, femoral artery catheterisation will be conducted in all cases

Immediately after induction of anesthesia :

Patients of group A will receive Dexmedetomidine which will be mixed with 0.9% saline to achieve a concentration of 4ug/ml which will continuously infused at a rate of 0.4 ug/kg/hr for 24 hours.

Patients of group B will receive an infusion of an equivalent volume of a 0.9% saline for the same duration

If hypotension occurred MAP will be maintained at 60-80 mm Hg using norepinephrine (maximum of 0.5ug/kg/min/) as necessary .

If bradycardia occurred low dose of atropine (0.01 mg\kg) can be given as necessary.

Institutionally standardised perioperative fluid and transfusion management will be conducted. Acute surgical bleeding or chest tube drainage will be compensated with allogeneic packed erythrocytes, depending on the haematocrit. Packed erythrocytes will be transfused when the haematocrit will be <20% during CPB or <25% otherwise. Fresh frozen plasma (FFP) and platelets will be transfused at the discretion of the attending anaesthesiologist and cardiac surgeon during surgery (Cho et al., 2016).

C.Postoperative settings:

After operation, if bleeding exceeded 200 m/h for 2 consecutive h, FFP, platelets, or both will be transfused if the international normalised ratio is greater than 1.3 or the platelet count is less than 50x103/ml. If oliguria occurred (urine output <1 ml/kg/h for 30 min), the volume status and appropriateness of haemodynamic values will be judged to determine the direction of treatment in all patients. Unless patients will be judged to have excessive circulating volume, three fluid boluses (200 ml of balanced crystalloid) will be administered. If the response will not be adequate 15 min after the third bolus or the patients' volume and haemodynamic status deemed appropriate, 5 mg furosemide will be administered intravenously, with repeated administrations every 30 min with escalating doses until the desired effect will be produced. Renal replacement therapy will be initiated if refractory oliguria, fluid overload, hyperkalaemia (>6.5 mEq\L) or rapidly increasing potassium levels, signs of uraemia, or metabolic acidosis (pH <7.1) occurred. Blood glucose levels will be adjusted according to the institutionally standardised insulin protocol .

Measurements and Data collection:

Demographic data as:

Age (years), sex (m/f), body, comorbidities, prior cardiac/aortic surgery

Introperative variables:

,Type of aortic surgey,duration of anaesthesia, CPB, Aortic cross clamp (ACC), and hypothermic circulatory arrest, fluid balance, , chest tube drainage, urine output, blood products transfusion, and the use of vasoconstrictors and inotropes for 48 h after surgery will be recorded after surgery. Haemodynamic data and laboratory data including serum creatinine, serum urea,serum electrolytes,haematocrit, white blood cell count, and C-reactive protein level will be serially assessed immediately after surgery and 12, 24 h, after surgery.

Outcomes:

The primary outcome: The primary outcome will be measurement of kidney function.AKI will be diagnosed based on the AKIN criteria: Stage 1 was defined as a serum creatinine increase ≥1.5-2-fold above baseline or ≥0.3 mg/dl or urine output <0.5 ml/kg/h for >6 h; stage 2 was defined as a creatinine increase >2-3-fold above baseline or urine output <0.5 ml/kg/h for >12 h; stage 3 was defined as a creatinine increase >3-fold above baseline or >4.0 mg/dl with an acute increase of 0.5 mg/dl, urine output <0.3 ml/kg/h for 24 h, or anuria for 12 h . Serum creatinine levels will be assessed before surgery, upon ICU arrival, at least once a day until postoperative day 5.

Secondary outcomes: For secondary outcomes, will be delirium, length of ICU stay, and inhospital mortality

Major morbidity end points:permenant stroke,hemostatic re-exploration,prolonged ventilator care> 48 hours

ELIGIBILITY:
Inclusion Criteria:

* ●Age: 20-70 yrs

  * Scheduled for aortic surgery under CPB

Exclusion Criteria:

* ●Patient refusal to participate

  * Congestive heart failure with a left ventricular ejection fraction <45%
  * Uncontrolled arrhythmia combined with unstable hemodynamics
  * Acute coronary syndrome.
  * Preoperative elevated kidney function (serum urea and serum creatinine). Use of ventricular assist devices

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
measurement of kidney function | Serum creatinine levels will beassessed before surgery, at least once a day until postoperative day 5
  AKI will be diagnosed based on the AKIN criteria: Stage 1 was defined as a serum creatinine increase ≥1.5-2-fold above baseline or ≥0.3 mg/dl or urine output <0.5 ml/kg/h for >6 h; stage 2 was defined as a creatinine increase >2-3-fold above baseline or urine output <0.5 ml/kg/h for >12 h; stage 3 was defined as a creatinine increase >3-fold above baseline or >4.0 mg/dl with an acute increase of 0.5 mg/dl, urine output <0.3 ml/kg/h for 24 h, or anuria for 12 h

SECONDARY OUTCOMES:
delirium | perioperative
  Delirium is a serious change in mental abilities. It results in confused thinking and a lack of awareness of someone's surroundings
inhospital mortality | perioperative
  the state of being subject to death

CONTACTS AND LOCATIONS:
Overall Officials: galal EL-KADY, MD, Study Director — Ain Shams University
Locations (1):
- AIN shams university, Cairo, Egypt, Egypt